CLINICAL TRIAL: NCT01093261
Title: Phase 3 Study of Hydrocortisone and Fludrocortisone in Glucocorticoid Insufficiency Related to Traumatic Brain Injury
Brief Title: Corticosteroid Therapy for Glucocorticoid Insufficiency Related to Traumatic Brain Injury
Acronym: Corti-TC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Collaborators: Société Française d'Anesthésie et de Réanimation (Other)
Responsible Party: Principal Investigator, Karim ASEHNOUNE, Asehnoune, Nantes University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BRD/10/01-L; SFAR (Other: Societe francaise d'Anesthesie Reanimation)
Record Dates: First submitted 2010-03-23; First posted 2010-03-25 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Traumatic Brain Injury; Trauma; Adrenal Insufficiency; Pneumonia
Keywords: trauma; trauma brain injury; multiple trauma; head trauma; hydrocortisone; fludrocortisone; glucocorticoid insufficiency related to ICU; adrenal Insufficiency; pneumonia; intensive care unit; shock; neurological recovery
MeSH Terms: conditions — Brain Injuries, Traumatic; Wounds and Injuries; Adrenal Insufficiency; Pneumonia; Multiple Trauma; Craniocerebral Trauma; Shock

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Hydrocortisone and fludrocortisone (Experimental): Patients with glucocorticoid insufficiency
  Interventions: Drug: Hydrocortisone Fludrocortisone
- Placebo (Placebo Comparator): Patients with glucocorticoid insufficiency
  Interventions: Drug: Placebo
- Controlled (No Intervention): Adapted glucocorticoid function

INTERVENTIONS:
Drug: Placebo — Placebo:
  continuous intra venous infusion of placebo n°1 for 10 days. enteral administration of placebo n°2 for 10 days.
  Arms: Placebo
Drug: Hydrocortisone Fludrocortisone — HYDROCORTISONE: 200 mg.day-1 for 7 days, 100 mg.day-1 on day 8 and 9, 50 mg on day-10 (continuous intravenous infusion) FLUDROCORTISONE: 50 microg.day-1 for 10 days (per os)
  Arms: Hydrocortisone and fludrocortisone

SUMMARY:
Traumatic brained injured (TBI) patients frequently suffered from glucocorticoid insufficiency that is associated with a raise in the rate of pneumonia.

In a placebo-controlled, multi-center, double-blinded trial, treatment of glucocorticoid insufficiency (hydrocortisone associated with fludrocortisone) will be assessed for prevention of post trauma pneumonia in a population of severe TBI patients.

DETAILED DESCRIPTION:
Treatment of glucocorticoid insufficiency in TBI patients remains controversial.

The purpose of this study is to determine whether hydrocortisone associated with fludrocortisone decreases rate of hospital-acquired pneumonia on day-28 in TBI patients with glucocorticoid insufficiency. Glucocorticoid function will be assessed by a corticotropin test (ACTH 0.25 mg). The study treatment will be started before reception of the results of these test. Patients with glucocorticoid insufficiency (basal cortisolemia < 15 mcg/dl or post ACTH raise < or = 9 mcg/dl) will be treated for 10 days. Patients with adapted glucocorticoid function will no longer be treated till the results of corticotropin test are known.

The primary end point will be rate of HAP on day-28 in patients with glucocorticoid insufficiency. Secondary endpoints will be neurological recovery (on day-28, -6 and -12), mortality (on day-28 and day-365), rate of other infections (on day-28), rate of organ failures (on day-28), mechanical ventilation weaning time, ICU length of stay.

In a double-blinded fashion (randomized on a 1:1 basis), 326 patients receive 200 mg intravenously for 10 days. After 7 days, treatment will be tapered with 100 mg given intravenously for days 8-9, then 50 mg for day 10, and then stopped.

All concomitant treatments, including antibiotics, fluids, vasopressors and ancillary therapies will be given at the discretion of the primary care physician. Evidence-based guidelines for the management of severe trauma brain injury (J Neurotrauma 2007; 24 Suppl 1, S1-106.) are encouraged to be followed. All institution are level I trauma center and university hospital.

Clinical assessments were performed twice a day in the ICU. When HAP was suspected after clinical examination, a new infiltrate was checked on a chest X-ray. The study protocol stated that antibiotic therapy should not be modified before a bacteriological sample was performed

All serious adverse events (SAE) which occur between days 0 and 28, which are unexpected and/or considered possibly or probably related to the study medication, must be documented and reported within 24 hours to the Safety and Efficacy Monitoring Committee. Non-serious adverse events will be listed on the case report form if they are unexpected and believed to be related to the study drug during days 0 to 14.

Specific adverse events which will be monitored closely because of their relationship to corticosteroids and trauma are: Use of corticosteroids, i.e. gastrointestinal bleeding and superinfection; hyperglycemia, hypernatremia, muscular weakness, etc.

In addition, substudies will include radiological assessment of hypothalamus and hypophyses,immune and neuro-endocrine interactions, post stress disorder assessment.

ELIGIBILITY:
Inclusion Criteria:

* Trauma brain injury (Glasgow score below 8 and lesion on scanner)
* Informed consent
* Time to inclusion inferior to 24 hours

Exclusion Criteria:

* Tetraplegia
* Administration of chronic corticosteroids in the last 6 months or acute steroid therapy (any dose) within 4 weeks (excluding inhaled steroids). Topical steroids are not exclusions
* Drug-induced immunosuppression, including chemotherapy or radiation therapy within 4 weeks before the study
* Antibiotherapy for active sepsis at the time of inclusion

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 336 (Actual)
Dates: Start 2010-08; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
rate of hospital acquired pneumonia | day-28
  Presence of at least two signs (body fever greater than 38°C; leukocytosis greater than 12000/ml or leukopenia below 4000/ml, purulent pulmonary secretions) associated with the appearance of a new infiltrate or modification of an existing infiltrate on chest-X-ray. Confirmation by a lower respiratory tract sample using a quantitative culture with a predefined positive threshold. Hospital-acquired pneumonia was defined as a pneumonia that occurs 48 hours after admission, which was not incubating at time of admission (Am J Respir Crit Care Med 2005; 171, 388-416).

SECONDARY OUTCOMES:
Neurological recovery | 1-year
  in adapated and insufficient glucocorticoid function (Glasgow Outcome Scale, Barthel index, MIF) (Ancillary study)
other infections | day-28
  Tracheobronchitis 1: Association of at least two signs (fever above 38.0°C, Leucocytosis above 12000/ml or purulent pulmonary secretions) with isolation of bacteria in a lower respiratory tract sample without modification of chest-X-Ray; Urinary tract infection : Fever above 38.2°C associated with leucocyturia (>10000/ml) and bacteriuria (>103 UFC/ml) without other infection; Bacteriemia : One positive blood culture (two positive blood cultures for Staphiloccocus coagulase negative); Surgical wound infection : sputum from surgical incision or scare dehiscence associated with fever.
Organ failures | day-28
  Acute Lung Injury or Acute Respiratory Distress Syndrom: PaO2/FiO2 below 300 with bilateral infiltrates on chest-X-ray without elevation of left atrial pressure; Acute kydney injury: oliguria (<0.3 ml/kg/hour for 24 hours or more) or raise in basal creatinemia of more than 300%; Myocardial insufficiency: indexed cardiac output below 2 l/min/m2; Hematologic insufficiency: platelet count below 50 000/ml; Hepatic insufficiency: bilirubinemia (<50 mmol.l-1) with a prothrombin (<40%), SOFA score (First week)
Length of ICU stay | 6 months
  in adapated and insufficient glucocorticoid function
Duration of mechanical ventilation support | 6 months
  in adapated and insufficient glucocorticoid function
Mortality from all causes | day-28
  in adapated and insufficient glucorticoid function
Mortality from all causes | 1 year
  in adapated and insufficient glucorticoid function
Time to amines withdrawal | day-28
Post traumatic stress disorder | 12 months
  Assessment of psychological status (ancillary study)
Glucocorticoid function | on day 11-12
  Short corticotropin test

CONTACTS AND LOCATIONS:
Overall Officials: Karim ASEHNOUNE, Study Chair — Nantes University Hospital; Antoine ROQUILLY, Principal Investigator — Nantes University Hospital; Pierre François Perrigault, Study Director — CHU de Montpellier; Pierre Albaladejo, Study Director — University Hospital, Grenoble; Marc Leonne, Study Director — CHU de Marseille; Olivier Langeron, Study Director — Assistance Publique Hopitaux de Paris
Locations (18):
- France (18):
  - University hospital, Amiens
  - University Hospital, Angers
  - University Hospital, Beaujon
  - University hospital, Bordeaux
  - University Hospital, Brest
  - Universtiy Hospital, Caen
  - University Hospital, Clermont-Ferrand
  - University hospital, Créteil
  - University Hospital, Créteil
  - University Hospital, Grenoble
  - University Hospital, Montpellier
  - University Hospital, Nantes
  - University Hospital, Nîmes
  - European Hospital Georges Pompidou, Paris
  - Saint Louis Hospital, Paris
  - University hospital, Poitiers
  - University Hospital, Strasbourg
  - University Hospital, Toulouse

REFERENCES:
- [Background] Asehnoune K, Roquilly A, Sebille V; Corti-TC trial group. Corticotherapy for traumatic brain-injured patients--the Corti-TC trial: study protocol for a randomized controlled trial. Trials. 2011 Oct 14;12:228. doi: 10.1186/1745-6215-12-228. PMID 21999663
- [Derived] Asehnoune K, Seguin P, Allary J, Feuillet F, Lasocki S, Cook F, Floch H, Chabanne R, Geeraerts T, Roger C, Perrigault PF, Hanouz JL, Lukaszewicz AC, Biais M, Boucheix P, Dahyot-Fizelier C, Capdevila X, Mahe PJ, Le Maguet P, Paugam-Burtz C, Gergaud S, Plaud B, Constantin JM, Malledant Y, Flet L, Sebille V, Roquilly A; Corti-TC Study Group. Hydrocortisone and fludrocortisone for prevention of hospital-acquired pneumonia in patients with severe traumatic brain injury (Corti-TC): a double-blind, multicentre phase 3, randomised placebo-controlled trial. Lancet Respir Med. 2014 Sep;2(9):706-16. doi: 10.1016/S2213-2600(14)70144-4. Epub 2014 Jul 24. PMID 25066331